CLINICAL TRIAL: NCT00141817
Title: A Multicenter, Randomized, Open Label, Single, and Multiple Dose Study of the Safety and Pharmacokinetics of 2 Dose Levels of Pantoprazole Sodium in Children Aged 1 Through 11 Years With Endoscopically Proven GERD
Brief Title: Study Evaluating Pantoprazole in Children With GERD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3001B3-334; B1791059
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2011-12-28 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2011-11

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastrointestinal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

INTERVENTIONS:
Drug: pantoprazole for approximately 9 weeks.

SUMMARY:
The purpose of this study is to characterize the PK profile, safety and tolerability of single and multiple doses of pantoprazole in children aged 1 through 11 years with endoscopically proven GERD.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopically proven GERD diagnosed within 6 months before study entry.
* Weight must be equal to or over 8.3 kg; for subjects 6 years or greater, weight must be equal to or under 25 kg

Exclusion Criteria:

* History of GI disorders, ie, unrepaired tracheal esophageal fistula, GI malabsorption, Eosinophilic esophagitis
* Subjects 6-11 years old unable to swallow tablets

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2005-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (22):
- United States (22):
  - Little Rock, Arkansas
  - Orange, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Pensacola, Florida
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - Detroit, Michigan
  - Flint, Michigan
  - Jackson, Mississippi
  - Kansas City, Missouri
  - New York, New York
  - Cincinnati, Ohio
  - Memphis, Tennessee
  - Temple, Texas
  - Salt Lake City, Utah
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Tammara BK, Sullivan JE, Adcock KG, Kierkus J, Giblin J, Rath N, Meng X, Maguire MK, Comer GM, Ward RM. Randomized, open-label, multicentre pharmacokinetic studies of two dose levels of pantoprazole granules in infants and children aged 1 month through <6 years with gastro-oesophageal reflux disease. Clin Pharmacokinet. 2011 Aug;50(8):541-50. doi: 10.2165/11591900-000000000-00000. PMID 21740077

RESULTS

PARTICIPANT FLOW:
Groups:
- Pantoprazole 0.6 mg/kg Spheroids: Pantoprazole 0.6 mg/kg Spheroids for Participants Aged <6 years
- Pantoprazole 1.2 mg/kg Spheroids: Pantoprazole 1.2 mg/kg Spheroids for Participants Aged <6 years
- Pantoprazole 0.6 mg/kg Tablets: Pantoprazole 0.6 mg/kg Tablets for Participants Aged >=6 years
- Pantoprazole 1.2 mg/kg Tablets: Pantoprazole 1.2 mg/kg Tablets for Participants Aged >=6 years
Period: Overall Study
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets
Started | 7 | 10 | 11 | 13
Completed | 6 | 10 | 10 | 13
Not Completed | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Parent request | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets | Total
Number analyzed (Participants) | 7 | 10 | 11 | 13 | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 3.86 (1.46) | 2.80 (1.55) | 8.55 (1.97) | 8.77 (1.09) | 6.41 (3.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 6 | 16
  Male | 5 | 6 | 7 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Predose (0 hour), and 0.5, 1, 2, 4, 6, 12 hours postdose
Population: Single-Dose Valid-for-Evaluation Population: Randomized participants who took 1 dose of pantoprazole and had at least 4 single-dose blood samples for pharmacokinetic (PK) analyses.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets
Number analyzed (Participants) | 3 | 7 | 10 | 13
nanogram per milliliter (ng/mL) | 136 (127) | 798 (729) | 1643 (1229) | 2067 (1320)

2. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Predose (0 hour), and 0.5, 1, 2, 4, 6, 12 hours postdose
Population: Single-Dose Valid-for-Evaluation Population. Participants analyzed=number of participants with available data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets
Number analyzed (Participants) | 3 | 7 | 10 | 12
hours | 1.45 (0.69) | 2.71 (1.25) | 2.08 (0.75) | 2.03 (0.74)

3. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]
Description: AUC (0-t)= Area under the plasma concentration versus time curve from time zero (predose) to time of last quantifiable concentration (0-t).
Time Frame: Predose (0 hour), and 0.5, 1, 2, 4, 6, 12 hours postdose
Population: Single-Dose Valid-for-Evaluation Population.
Measure: Mean (Standard Deviation); unit: nanogram hour per milliliter (ng*h/mL)
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets
Number analyzed (Participants) | 3 | 7 | 10 | 13
nanogram hour per milliliter (ng*h/mL) | 208.96 (197.54) | 2273.96 (1885.68) | 2448.61 (2007.21) | 3190.96 (2137.91)

4. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (predose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: Predose (0 hour), and 0.5, 1, 2, 4, 6, 12 hours postdose
Population: Single-Dose Valid-for-Evaluation Population. Participants analyzed=number of participants with available data.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets
Number analyzed (Participants) | 3 | 7 | 10 | 11
ng*h/mL | 293.29 (146.41) | 2448.08 (2170.48) | 2497.13 (2099.64) | 3782.49 (1837.42)

5. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Predose (0 hour), and 0.5, 1, 2, 4, 6, 12 hours postdose
Population: Single-Dose Valid-for-Evaluation Population. Participants analyzed=number of participants with available data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets
Number analyzed (Participants) | 3 | 7 | 10 | 11
hours | 5.34 (7.39) | 1.68 (0.64) | 0.77 (0.22) | 0.70 (0.16)

6. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Predose (0 hour), and 0.5, 1, 2, 4, 6, 12 hours postdose
Population: Single-Dose Valid-for-Evaluation Population. Participants analyzed=number of participants with available data.
Measure: Mean (Standard Deviation); unit: liter per hour per kilogram (L/h/kg)
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets
Number analyzed (Participants) | 3 | 7 | 10 | 11
liter per hour per kilogram (L/h/kg) | 2.08 (1.27) | 1.28 (1.16) | 0.41 (0.30) | 0.40 (0.22)

7. Primary Outcome: Terminal-Phase Volume of Distribution (Vz/F)
Description: Vz/F was calculated as the ratio of clearance (CL) to terminal disposition rate constant (λz).
Time Frame: Predose (0 hour), and 0.5, 1, 2, 4, 6, 12 hours postdose
Population: Single-Dose Valid-for-Evaluation Population. Participants analyzed=number of participants with available data.
Measure: Mean (Standard Deviation); unit: liter per kilogram (L/kg)
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets
Number analyzed (Participants) | 3 | 7 | 10 | 11
liter per kilogram (L/kg) | 12.22 (14.68) | 2.89 (2.92) | 0.43 (0.30) | 0.40 (0.27)

8. Primary Outcome: Plasma Concentrations After Multiple Doses
Time Frame: Hours 2 and 4 on Day 7
Population: Multiple-Dose Valid-for-Evaluation Population: Randomized participants who had concentration evaluations of pantoprazole either at 2 hours or at 4 hours after single dose and after at least 5 consecutive doses. n=participants who had data available at that specific time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets
Number analyzed (Participants) | 6 | 8 | 10 | 13
ng/mL
  Hour 2 on Day 7 (n=5, 8, 10, 13) | 212.30 (222.08) | 486.49 (605.22) | 592.32 (914.57) | 2337.89 (1817.78)
  Hour 4 on Day 7 (n=6, 8, 10, 13) | 503.25 (1087.91) | 207.23 (211.92) | 123.83 (163.78) | 200.78 (209.81)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Pantoprazole 0.6 mg/kg Spheroids | Pantoprazole 1.2 mg/kg Spheroids | Pantoprazole 0.6 mg/kg Tablets | Pantoprazole 1.2 mg/kg Tablets
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10 | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 4/7 | 7/10 | 9/11 | 7/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pantoprazole 0.6 mg/kg Spheroids (N=7) | Pantoprazole 1.2 mg/kg Spheroids (N=10) | Pantoprazole 0.6 mg/kg Tablets (N=11) | Pantoprazole 1.2 mg/kg Tablets (N=13)
Abdominal pain (General disorders) | 1 | 1 | 3 | 1
Accidental injury (General disorders) | 1 | 1 | 1 | 1
Fever (General disorders) | 0 | 1 | 1 | 1
Hypotension (Cardiac disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Creatine phosphokinase increased (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Thirst (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Weight loss (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Abnormal/changed behavior (Nervous system disorders) | 1 | 0 | 0 | 0
Cough increased (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Otitis media (Ear and labyrinth disorders) | 0 | 1 | 2 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1 | 0 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Headache (General disorders) | 0 | 0 | 1 | 2
Injection site hemorrhage (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hyperlipemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.